CLINICAL TRIAL: NCT05389826
Title: mHealth System for the Self-control of Hyperphosphatemia in Patients With CKD.
Brief Title: mHealth for Phosphorus Management in CKD.
Acronym: PHOSFO_OK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, MIGUEL HUESO VAL, Principal Investigator; Staff member of Nephrology Department, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR291/21
Record Dates: First submitted 2022-05-13; First posted 2022-05-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Dialysis Related Complication
Keywords: mHealth; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Intervention Model Description: Pilot study involving cases and controls. Fifty outpatient patients with stage 4-5 CKD, including those on dialysis will be included. Twenty-five patients will be followed with the developed mobile web app, while another twenty-five patients will be treated according to the current clinical practice. Patients will be randomized blindly 1:1 to the study group or to the control group. The randomization technique consists of consecutively numbered sealed envelopes on which the signed group is written.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth App group (Experimental): Patients will be followed with the developed mobile web app,
  Interventions: Device: mHealth App
- Control (No Intervention): Patients will be treated according to the current clinical practice.

INTERVENTIONS:
Device: mHealth App — We will compare the degree of improvement in phosphate control with respect to baseline values and report any adverse event. Nephrologist will use a web management system to provide results of phosphorus levels and medical recommendations to the patient, mediated by a cloud IT environment. In addition, patients will receive alerts, suggestions, and general information. They will also be able to communicate with nephrologists and interact with their corresponding group of fellow patients.
  Arms: mHealth App group

SUMMARY:
The project aims to generate an mHealth environment in which CKD patients are empowered in terms of the self-management of their hyperphosphatemia pathology, while under medical supervision. Such environment will allow nephrologists to inform patients beyond their traditional point-of-care and will allow patients to provide feedback on their condition in a timely manner that benefits the CKD collective. In this way we delve in a technological area that has been argued that remains underutilized within nephrology (1) and that should be perceived as an opportunity for CKD (2). In our work, we will build from recent related efforts in the control of hyperphosphatemia (3).

DETAILED DESCRIPTION:
The working hypotheses are listed as follows:

1. Hyperphosphatemia is an important problem in the CKD realm, but difficult to manage because patients are often not aware of its importance. In addition, current clinical practice does not allow nephrologists to evaluate the patient's real understanding of their recommendations.
2. The patient could benefit from a smartphone-based interactive virtual assistant tool: an integrated personalized management system to achieve a form of participatory, personalized, predictive and preventive medicine in the specific domain of a pathology associated to CKD.
3. The combination of a flexible information channel with an interactive data visualization tool on mobile devices can be a most intuitive way to communicate with the patient, particularly if it allows comparison with other patients in similar situation. Additionally, data visualization can assist nephrologists in the clinical management of patients.

Primary Objective:

1-Analysis of the superiority of a Medical Mobile Application for Patient Support to educate CKD patients on how to self-manage their phosphate levels versus standard of care in lowering serum phosphorus by assessing changes in serum phosphorus comparing baseline with 6-months follow-up.

Secondary Objectives:

1. Adherence to treatment with phosphate binders.
2. Impact in Quality of Life of patients with CKD.
3. Satisfaction of such a tool.

ELIGIBILITY:
Inclusion Criteria:

1- Eligible patients will be stage 4-5 CKD patients, including end-stage renal disease (ESRD) on dialysis, aged >18 with hyperphosphatemia (serum phosphorus concentration >1.94 mmol/L) and stable dose of phosphate binders for >1 month before screening.

Exclusion Criteria:

1. Patients with intact parathyroid hormone concentration >800 ng/l (88 pmol/l) or if parathyroidectomy will be planned or expected.
2. Patients with significant gastro-intestinal (GI) or hepatic disorders.
3. Patients with major GI surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Analysis of the superiority of mobile-app and benchmarking versus standard of care in lowering serum phosphorus | 6-months follow-up
  Reduction of serum phosphorus by more than 0.5 mmol/L versus the standard of care testing.

SECONDARY OUTCOMES:
Adherence to phosphate binder's use and reduction in their use. | 6-months follow-up
  The ratio of current phosphate binders that the patient is swallowing compared to the number prescribed.
Quality of life improvement | 6-months follow-up
  Health-related quality of life (HRQoL) will be assessed with the Short-Form 12 questionnaire (SF-12).
Patient's and healthcare professionals' satisfaction with mobile health app to ensure its usability and promote patient retention | 6-months follow-up
  Satisfaction of patients will be assessed with the quality of care satisfaction in outpatient consultation questionnaire (EQS-C).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Reporting the study design
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months
Access Criteria: Publication

REFERENCES:
- [Background] Stauss M, Dhaygude A, Ponnusamy A, Myers M, Woywodt A. Remote digital urinalysis with smartphone technology as part of remote management of glomerular disease during the SARS-CoV-2 virus pandemic: single-centre experience in 25 patients. Clin Kidney J. 2021 Dec 21;15(5):903-911. doi: 10.1093/ckj/sfab286. eCollection 2022 May. PMID 35498887
- [Background] Topf JM, Hiremath S. Got CKD? There's an App for That! Clin J Am Soc Nephrol. 2019 Apr 5;14(4):491-492. doi: 10.2215/CJN.02350219. Epub 2019 Mar 21. No abstract available. PMID 30898874
- [Background] Chiang YC, Chang YP, Lin SC, Lin C, Hsu PH, Hsu YJ, Wu TJ. Effects of Individualized Dietary Phosphate Control Program With a Smartphone Application in Hemodialysis Patients in Taiwan. Biol Res Nurs. 2021 Jul;23(3):375-381. doi: 10.1177/1099800420975504. Epub 2020 Nov 28. PMID 33251815